CLINICAL TRIAL: NCT05558215
Title: Remote Online Administration of Otago Exercise Program for Individuals With Dementia and Their Care Partners: A Feasibility Study
Brief Title: Remote Balance Training for Individuals With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marymount University (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Julie Ries, Professor of Physical Therapy, Research Fellow of Center for Optimal Aging, Marymount University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ARDRAF 22-3
Record Dates: First submitted 2022-09-19; First posted 2022-09-28 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Dementia
Keywords: Balance; Exercise; Dementia
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single group clinical trial with single arm to assess feasibility of remote administration of balance training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Otago Exercise Program (Experimental): Individuals with dementia will participate in Otago Exercise Program in their home using video recordings and with safety oversight by their trained care partners.
  Interventions: Other: Otago Exercise Program

INTERVENTIONS:
Other: Otago Exercise Program — The Otago Exercise Program (OEP) is a CDC endorsed evidence-based falls prevention program for older adults. It has not been well studied with individuals with dementia. It is comprised of a brief "warm up"/flexibility series, lower extremity strengthening, and balance exercises. The same menu of exercises is used for all participants, but exercises are progressed based upon individual performance. For the purposes of this study, three 25-minute video recorded versions of OEP will be rotated for use, all of which include brief flexibility activities, strengthening, and balance exercises. Strengthening exercises will be limited to body weight resistance for ease of instruction, safety, and consistency. Balance exercises involve changes in base of support in static and dynamic contexts, with challenge progressively increased by decreasing arm support during training (from 2-hands, to 1-hand, to no hands).
  Other Names: Modified Otago Exercise Program

SUMMARY:
Individuals with dementia (IwDs) fall more and are more seriously injured in falls than their age-matched, cognitively intact peers. An accessible and sustainable fall prevention program would be of great value. Using remote technology has become commonplace during the COVID-19 pandemic, and Marymount University's new Center for Optimal Aging plans to use this technology to bring a web-based version of a well-established and accepted evidence-based fall prevention intervention, the Otago Exercise Program, into the homes of IwDs and their care partners. Care partners will be trained in the home for safety and oversight of their exercising partner with dementia. Dyads of IwD and care partners will access the online exercise program through an online Learning Management System (Canvas) three times per week which tracks their access to exercise videos. Once per week, exercise will take place in a Zoom format with a small cohort of other dyads, supervised by a research team member, and the other two times will be independent access of exercise videos. The purpose of this study is to determine the viability of remote administration of the Otago Exercise Program by assessing program functionality, utility, and effectiveness. Feasibility will be evaluated by using components of the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance). The results will guide and inform adaptations of future remote training efforts for IwD, with implications at the individual, family, and societal levels.

DETAILED DESCRIPTION:
Methodology Overview:

This 16-week prospective study will examine feasibility of remotely administered Otago Exercise Program (OEP) for Individuals with Dementia (IwD) supervised by their care partners (n=24 dyads) using select components of the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance). Specifically, data on program adherence, system usability, enjoyment, and adverse events will inform the ability of Marymount Center for Optimal Aging to work with partners to Adopt and Implement this programming for the older adult community. Additionally, this within-subject design study will assess measures of balance, mobility, falls, cognition, & confidence to assess preliminary data on Effectiveness, should the program be feasible. Finally, Reach will be evaluated by comparing demographic data of participants recruited as compared to the target local community, which is broadly diverse in terms of age, race, ethnicity, economic status, health status, culture, and language.

Existing studies demonstrate that home based exercise for IwD with care partners are feasible and safe, providing there is careful orientation to safety measures and continued support and follow up over the course of the study. Inclusion/exclusion criteria are designed to avoid inclusion of very high risk fallers (i.e., use of assistive device).

All assessments will be performed in the participant's home with oversight by a licensed physical therapist (PT) with geriatric expertise. A PT/PT student team will be assigned to each dyad for the duration of the study and the team will have regular contact with the dyad to direct activities, discuss questions and concerns, and provide support over the initial 8-weeks of the study, and waning contact over the final 8-weeks of the study. Students will be vetted and trained by the PTs. A detailed procedures manual describing all testing, remote exercise administration, and data collection procedures will be followed by all research team members.

After an enrollment visit and consent, pre-test assessment, and education/safety training for home exercise (Week 0), IwD with care-partner supervision will participate in remote OEP (3x/week x 8 weeks) with 1x/week synchronous/real time with an online research team instructor and small group (<3) of other dyads. The other sessions (2x/wk) will be carried out independently by dyads using pre-recorded videos of exercises without live instruction. Following completion of the 8-wk OEP, immediate post-testing (Week 8) will occur.

For Weeks 9-16, dyads will be encouraged to continue with OEP videos 3x/week, but there will no longer be synchronous/research team supervised sessions. There will be continued weekly opportunity to meet with other dyad participants via Zoom. Study personnel will contact dyads via phone/email/zoom (per participant preference) to provide encouragement and answer questions. The frequency of contact will fade over Weeks 9-16: Weekly for Weeks 9-10; every other week for Weeks 11-14; and only as requested for Weeks 15-16 (i.e., when the participant initiates contact). Delayed post-testing will occur following Week 16.

Specific Procedures and Intervention:

Enrollment Visit: An Enrollment visit will be scheduled after phone screening which will include: (1) Care partner screening to assure ability to safely oversee exercise program; (2) Answer any questions & procure signed consent; (3) Intake demographic & medical data; (4) Education re: location & set up for safe exercising; and (5) Introduction to remote platforms for use during study.

Home Visit 1 @ Week 0: Includes: (1) Data collection of outcome measures for pre-OEP; (2) Review Canvas & Zoom platform access; (3) Review education re: location & set-up for safe exercising; and (4) Provide OEP manual and calendar/diary.

OEP Intervention (remote supervision 1x/week, independent dyad exercise 2x/week) Weeks 0-8: The research team will work with dyads (during preparation, synchronous sessions & weekly check-ins) to assure safety as the top priority and to encourage maximal participant challenge during exercise sessions. OEP will be administered via a web-based learning management system (Canvas). The Canvas site set-up will be simple, with two links, one for the synchronous classes (1x/week) and one for asynchronous classes (2x/week). Synchronous classes (3-4 dyads) will be carried out using a video conferencing application (Zoom) with oversight by a research team member. A video of OEP exercise will run on the shared screen throughout the exercise activity. The videos instruct safe progression of exercises. Participant dyads will access asynchronous online OEP sessions twice per week independently with videos accessed through Canvas. Participant dyads will receive weekly check-in calls/emails/Zoom meetings (based upon participant preference) from their PT / student team to stay connected, share falls diary data, and have an opportunity to ask questions.

Home Visit 2 @ Week 8: Includes: (1) Data collection of outcome measures for post-OEP-1; and (2) Data collection for feasibility measures-1 with dyads.

OEP Intervention (independent dyad exercise 3x/wk) Weeks 9-16: Participants are encouraged to continue to perform OEP 3x/wk without direct supervision by research staff. Fading frequency of check-ins over the course of weeks 9-16, but continued opportunity and encouragement to communicate on Zoom with other participant dyads and discuss OEP experience. These opportunities will occur weekly at the shared Zoom link at agreed upon times for the small group of dyads that had exercised together during weeks 0-8.

Home Visit 3 @ Week 16: Final home visit includes: (1) Data collection of outcome measures for post-OEP-2; and (2) Data collection for feasibility measures-2 with dyads.

Data Management & Analysis:

All research team members, including students, will be educated in research ethics, participant privacy, and data confidentiality, and will act accordingly in the context of data management. Data collection in the home will occur using password protected tablet with electronic forms. Participants will be assigned a Research ID number which will be associated with their data. Research ID numbers associated with direct identifiers will be stored separately from collected data, and personal health information will be kept to a minimum. Data used for analysis will be de-identified. Data shared in publications or presentations will be presented in aggregate or summary form such that no individuals are identifiable. Publication / presentation of data shall be consistent with normal scientific practices.

Feasibility data will be evaluated with some measures compared to a priori thresholds and others evaluated descriptively. Adherence data will be compared to mean adherence rates (proportion of classes attended) for falls prevention programs for older adults, which is 66%. System Usability Scale (SUS) scores will be assessed relative to a priori target score of >65, as modeled by others using remote technology with a similar population. Adverse events, PACES-8 (enjoyment) and BSFC (caregiver burden) data will not have a priori thresholds, but will be descriptively presented and compared to other studies. Functional tests (30sCST, TUG) will be assessed with paired t-tests to determine immediate intervention impact (Week 0 vs Week 8), and with Repeated-measures ANOVA across 3 testing sessions (Week 0, Week 8, Week 16); non-parametric 4-stage balance test will be evaluated with Wilcoxon test (Week 0 vs Week 8) and with Friedman test across 3 sessions, and with attention to the identified threshold score (marking high to lower fall risk).

ELIGIBILITY:
Inclusion Criteria for IwD:

* English-speaking, community-dwelling adults >60 years old
* Physician's confirmed diagnosis of mild to moderate dementia
* Medical stability (indicates absence of all medical conditions listed in exclusion criteria and effective medical management of medical issues [e.g., hypertension is managed by medication]).
* Ability to walk indoors without assistive device or physical assistance of another person
* Ability to follow one-step commands
* A committed care provider / person responsible willing to supervise exercise sessions 3x/wk

Exclusion Criteria for IwD:

* Use of assistive device or furniture for indoor walking
* Advanced dementia
* Acute / severe psychiatric condition
* Unstable or limiting systemic pathology (e.g., cardiac, pulmonary, metabolic, orthopedic, neurologic)
* Recent (within 6 months) major surgical intervention (for any reason) or treatment for cancer
* Neurological diagnosis/condition with residual deficit (e.g., stroke, Parkinson's Disease).

Inclusion Criteria for Care Partner:

* English speaking
* Cognitively & physically capable of providing safety oversight to IwD during balance training program
* Has computer /tablet with internet access for use in the home of the IwD
* Committed to overseeing IwD for exercise program 3x/week
* Willing to maintain fall diary and participate in providing data for feasibility measures.

Exclusion Criteria for Care Partner:

* Uses assistive device for mobility
* General health and/or wellness prohibits oversight of IwD during exercises
* Inability to master technology required for project

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender data collected will be participant's self-identified gender.
Enrollment: 18 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Change over time (pre-intervention, immediate post-intervention, delayed post-intervention) in 4-Stage Balance Test (4-SBT) | Assessed at Weeks 0, 8, and 16
  The participant will stand with feet in four different positions and be timed for up to 10 seconds in each position. The positions are: (1) feet side by side, (2) staggered stance with feet next to each other, (3) one foot in front of the other, and (4) standing on one foot.
Change over time (pre-intervention, immediate post-intervention, delayed post-intervention) in 30-second Sit to Stand (30s STS) | Assessed at Weeks 0, 8, and 16
  The number of stands completed in 30 seconds without use of arms from a standard kitchen or dining room chair (standard test is with 17-inch seat to floor height).
Change over time (immediate post-intervention, delayed post-intervention) in Adherence / Participation | Assessed at Weeks 8 and 16
  Measured by attendance & participation at synchronous sessions and by number of "views" recorded through Canvas website for asynchronous sessions.
Change over time (immediate post-intervention, delayed post-intervention) in System Usability Scale (SUS) | Assessed at Weeks 8 and 16
  SUS is a 10-item Likert survey and scores are between 0-100 with higher scores representing better usability.

SECONDARY OUTCOMES:
Change over time (pre-intervention, immediate post-intervention, delayed post-intervention) in Timed Up and Go (TUG) | Assessed at Weeks 0, 8, and 16
  Measures time taken to stand, walk 3 meters, turn and walk back, and sit.
Change over time (pre-intervention, immediate post-intervention, delayed post-intervention) in Short Falls Efficacy Scale-International (Short FES-I) | Assessed at Weeks 0, 8, and 16
  Short FES-I is a 7-item Likert scale measure of subjective fear/concern about falling. Scores range from 7 to 28 with higher scores representing MORE concern about falling (i.e., worse outcome).
Change over time (pre-intervention, immediate post-intervention, delayed post-intervention) in Burden Scale for Family Caregivers-Short Version (BSFC). | Assessed at Weeks 0, 8 and 16
  BSFC is a 10-item Likert scale measure of the subjective impact of providing care on the care provider. Scores range from 0 to 84 with higher scores representing MORE perceived burden by care provider (i.e., worse outcome).
Change over time (pre-intervention and delayed post-intervention) in Montreal Cognitive Assessment (MoCA). | Assessed at Weeks 0 and 16
  Brief (30-item) cognitive screening tool that includes multiple domains of cognitive functioning. Scores range from 0-30 with higher scores representing higher levels of cognitive functioning (i.e., better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Heyn, PhD, Study Director — Marymount University Center for Optimal Aging; Rita Wong, EdD, Study Director — Marymount University
Locations (1):
- Marymount University, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Suttanon P, Hill KD, Said CM, Williams SB, Byrne KN, LoGiudice D, Lautenschlager NT, Dodd KJ. Feasibility, safety and preliminary evidence of the effectiveness of a home-based exercise programme for older people with Alzheimer's disease: a pilot randomized controlled trial. Clin Rehabil. 2013 May;27(5):427-38. doi: 10.1177/0269215512460877. Epub 2012 Nov 1. PMID 23117349
- [Background] Taylor ME, Close JCT, Lord SR, Kurrle SE, Webster L, Savage R, Delbaere K. Pilot feasibility study of a home-based fall prevention exercise program (StandingTall) delivered through a tablet computer (iPad) in older people with dementia. Australas J Ageing. 2020 Sep;39(3):e278-e287. doi: 10.1111/ajag.12717. Epub 2019 Sep 19. PMID 31538401
- [Background] Osho O, Owoeye O, Armijo-Olivo S. Adherence and Attrition in Fall Prevention Exercise Programs for Community-Dwelling Older Adults: A Systematic Review and Meta-Analysis. J Aging Phys Act. 2018 Apr 1;26(2):304-326. doi: 10.1123/japa.2016-0326. Epub 2018 Apr 23. PMID 28771111